CLINICAL TRIAL: NCT03852940
Title: Impact of Early Enteral vs. Parenteral Nutrition on Preservation of Gut Mucosa Integrity in Patients Requiring Mechanical Ventilation and Catecholamines: an Ancillary Study of the NUTRIREA2 Trial (NCT01802099)
Brief Title: Impact of Early Enteral vs. Parenteral Nutrition on Preservation of Gut Mucosa Integrity in Patients Requiring Mechanical Ventilation and Catecholamine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data Safety and Monitoring Board 's request
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Ministry of Health, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHD085-12
Record Dates: First submitted 2017-07-18; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2017-07

CONDITIONS: Acute Respiratory Failure; Shock
Keywords: vasoactive drug; mechanical ventilation; early enteral nutrition; intensive care unit; early parenteral nutrition; critical care medicine; nosocomial infection; mortality; shock
MeSH Terms: conditions — Shock; Hyperphagia; Cross Infection | interventions — Parenteral Nutrition; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parenteral nutrition (Other): Patients will receive parenteral nutrition during the first week of mechanical ventilation. After Day 3, the parenteral route may be switched to the enteral route if shock resolve (vasoactive drug stopped since 24 hours and serum lactate level < 2 mmol/l). After Day 7, all patients will be fed via the enteral route.
  Interventions: Other: Parenteral nutrition
- Enteral nutrition (Other): Patients will receive nutrition only via the enteral route during the firs week of invasive mechanical ventilation.
  Interventions: Other: Enteral Nutrition

INTERVENTIONS:
Other: Parenteral nutrition
  Other Names: Intravenous nutrition; intravenous feeding
  Arms: Parenteral nutrition
Other: Enteral Nutrition
  Other Names: Enteral feeding
  Arms: Enteral nutrition

SUMMARY:
To demonstrate that a strategy involving early first-line enteral nutrition is associated with improved preservation of gut mucosa integrity, as assessed based on the plasma citrulline level at H72, compared to a strategy involving early first-line parenteral nutrition

DETAILED DESCRIPTION:
Published data suggest that enteral nutrition may be associated with improved preservation of the gut lymphoid tissues and gut immune function, as well as with decreased gut mucosa permeability, thereby diminishing the risk of organ failure. Citrulline is an amino acid produced from glutamine by small-bowel enterocytes. Plasma citrulline levels reflect functional enterocyte mass. Intestinal fatty acid-binding protein (I-FABP, also known as FABP2) is a small protein found in the cytosol of small-bowel enterocytes. Plasma I-FABP is normally undetectable and, when elevated, constitutes a reliable marker for enterocyte damage. The hypothesis underlying this ancillary study is that first-line enteral nutrition is associated with improved gut mucosa integrity and function compared to parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation expected to be required more than 48 hours
* Nutrition started within 24 hours after initiation of endotracheal mechanical ventilation
* Treatment with vasoactive drug administered via a central venous catheter
* Age over 18 years
* Signed information

Exclusion Criteria:

* Abdominal surgery within 1 month before inclusion
* History of esophageal, gastric, duodenal or pancreatic surgery
* Bleeding from the esophagus, stomach or bowel
* enteral nutrition via gastrostomy or jejunostomy
* pregnancy
* Treatment-limitation decisions
* Current inclusion in a trial on comparison between enteral and parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2015-07-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Plasma citrulline level | 72 hours

SECONDARY OUTCOMES:
SOFA score | first week
plasma levels of citrulline | Day 0, Day 3, Day 8
I-FABP | Day 0, Day 3, Day 8
proportion of patients whose plasma I-FABP is ≥100 pg/mL | Day 0, Day 3, Day 8
proportion of patients whose plasma citrulline is ≤10 μL/L | Day 0, Day 3, Day 8
mean plasma I-FABP | Day 0, Day 3, Day 8
mean plasma citrulline | Day 0, Day 3, Day 8
proportion of patients with at least one episode of bacteremia | until discharge from ICU (average: 10 days)
proportion of patients with at least one episode of gastrointestinal intolerance | until discharge from ICU (average: 10 days)
proportion of patients with at least one episode of diarrhea | until discharge from ICU (average: 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jean REIGNIER, MD, PhD, Principal Investigator — CHD Vendee
Locations (6):
- France (6):
  - CHU Amiens, Amiens
  - Centre hospitalier d'Annecy, Annecy
  - CH de Dieppe, Dieppe
  - CHU Lille, Lille
  - CHU Saint Louis, Paris
  - CHU Tours, Tours